CLINICAL TRIAL: NCT00828503
Title: Certican® (Everolimus) Against Cytomegalovirus Disease in Renal Transplant Patients
Acronym: Certi-CMV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marcus Saemann (Other)
Responsible Party: Sponsor-Investigator, Marcus Saemann, Ass. Prof. Dr. Marcus Säemann, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2008-004745-28
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Cytomegalovirus Disease
Keywords: Certi-CMV; immunosuppressive switch (to Certican); renal transplant
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Everolimus; Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Certican + Valganciclovir (Active Comparator): Valganciclovir will be administered and Certican (everolimus) will be added as immunosuppression
  Interventions: Drug: Certican (everolimus) + valganciclovir
- 2 Valganciclovir alone (Active Comparator): Valganciclovir will be added alone.
  Interventions: Drug: Valganciclovir

INTERVENTIONS:
Drug: Certican (everolimus) + valganciclovir — Oral MED 1: Certican® initial dose: 1,5-3 mg day target trough level: 3-8 ng/mL (first levels will be performed after 3 days and then adjusted until - according to the judgement of the clinical investigator - a stable degree of immunosuppression is reached; thereafter Certican® trough levels will be performed at the scheduled appointments)
  MED 2: Valganciclovir (or ganciclovir) will be administered in addition to Certican (valganciclovir: 450 mg twice daily, ganciclovir 5 mg/kg i.v. twice daily)
  Arms: 1 Certican + Valganciclovir
Drug: Valganciclovir — Valganciclovir (or ganciclovir) will be administered alone (valganciclovir: 450 mg twice daily, ganciclovir 5 mg/kg i.v. twice daily)
  Arms: 2 Valganciclovir alone

SUMMARY:
A prospective, randomized safety and efficacy study of Certican® as add-on therapy against CMV disease in renal transplant recipients

OBJECTIVES:

Primary Objective:

To demonstrate efficacy of Certican® as add-on therapy against CMV disease in comparison to either valcyte® (valganciclovir) or cymevene® (ganciclovir) alone, evaluated by quantitative measurement of CMV-DNA with PCR from the blood (qCMV-PCR)

Secondary Objectives:

To assess safety and tolerability of Certican® in patients with CMV- disease To study the effects of Certican® treatment on quality of life

DETAILED DESCRIPTION:
DESIGN / PHASE Prospective, single-center, randomized, parallel group, controlled, phase II study.

PATIENTS / GROUPS 40 patients in 2 groups 20 patients per group Randomization ratio 1:1, no stratification

INVESTIGATIONAL DRUG Oral MED 1: Certican® initial dose: 1,5-3 mg day target trough level: 3-8 ng/mL (first levels will be performed after 3 days and then adjusted until - according to the judgment of the clinical investigator - a stable degree of immunosuppression is reached; thereafter Certican® trough levels will be performed at the scheduled appointments)

COMPARATIVE DRUG No therapy (add-on design

CONCOMITANT MEDICATION Allowed The concomitant immunosuppressive medication will be adjusted to the additional administration of Certican®. For example, if the patient already receives cyclosporine A or tacrolimus, this will be adjusted, according to the current recommendations4 at the judgment of the clinical investigator

TOLERABILITY / SAFETY ENDPOINTS:

Rejection Hematocrit Platelet count WBC count Wound healing disorders Blood lipids (cholesterol, triglycerides) Infections (other than CMV)

PHARMACOKINETIC / PHARMACODYNAMIC ENDPOINTS Certican® (everolimus) trough levels

STATISTICAL METHODOLOGY Primary Endpoint: CMV-load (copies/mL)

Null and alternative hypotheses:

H0 Treatment with Certican® (everolimus) in combination with valcyte® (valganciclovir) or cymevene® (ganciclovir) is equal to valcyte® (valganciclovir) or cymevene® (ganciclovir) alone in reducing the CMV-load in renal transplant patients with CMV-disease H1: Treatment with Certican® (everolimus) in combination with valcyte® (valganciclovir) or cymevene® (ganciclovir) is superior to valcyte® (valganciclovir) or cymevene® (ganciclovir) in reducing CMV load (copies/mL) in renal transplant patients with CMV-disease Type-I and -II errors - power. α=0.05 ß=0.2 (power 0.8) Statistical methodology ANOVA of repeated measures (CMV-copies/mL), one-sided t-test of CMV load at distinct time-points, one-sided t-test of the time (in weeks) until CMV-load reaches ≤600 copies/mL Sample size calculation Based on a one-sided testing and a σ of 0.2 in relative changes of CMV-copies, an α=0.05 And a ß=0.2 a sample size of 20 patients per group was determined. Main analysis set Per-protocol (efficacy) and intention to treat (ITT) for safety Other endpoints Bonferroni corrected t-tests will be performed for CMV-copies/mL at each time point of the follow-up period. The time to copies ≤ 600 will also be analyzed by a t-test. All other secondary endpoints and subgroup analysis will be performed in explorative intention (descriptive statistics).

ELIGIBILITY:
Inclusion Criteria:

* CMV-disease after renal transplantation, i.e.,(1.) CMV present in the blood, and (2.) one of the following symptoms (for viral syndrome, from the American Society of Transplantation recommendations for use in clinical trials1):

  * body temperature ≥ 38°C
  * new or increased significant malaise
  * leucopenia (< 3500/mL)
  * atypical lymphocytosis ≥ 5%
  * thrombocytopenia (platelets < 100.000/mL)
* no other cause of symptoms/signs identified
* informed consent of the patient

Exclusion Criteria:

* patients with a known hypersensitivity to everolimus, sirolimus or any of the excipients
* administration of strong CYP3A4 Inhibitors (e.g. ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin) and inducers (rifampicin), unless the benefit outweighs the risk, according to the judgment of the clinical investigator
* acute rejection episodes in the first 3 months after renal transplantation
* active hepatitis in the previous month
* Significant proteinuria (> 0.8g/24h Urine)
* hepatic impairment, according to the criteria defined by Bénichou et al.2: a singular elevation of GPT or conjugated bilirubin to a value twice above the normal level, or a combined elevation of GOT, AP, and total bilirubin, given that at least one parameter is twice above the normal level
* hematocrit < 25%
* any significant wound healing disorder (anamnestic)
* blood white blood cell (WBC) count < 3000/mL
* platelets < 50.000/mL
* severe dyslipidemia (cholesterol >300mg/dL, triglycerides > 350mg/dL)
* uncontrolled hypertension (continuous episodes of hypertension above 140/90 (WHO classification and American Society of Transplantation recommendations 3) despite adequate hypertensive therapy)
* uncontrolled hyperuricemia (uric acid > 8mg/dL)
* pregnancy
* any immunosuppressive protocol which does not allow the addition of Certican®, according to the judgment of the clinical investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
relative changes in CMV-load (copies/mL), as determined by qCMV-PCR from whole blood throughout the observational period | 2 years

SECONDARY OUTCOMES:
CMV-load (copies/mL) after 1-8 weeks, in months 3, 4, 6 and 12; Time (in weeks) until the CMV-load reaches ≤600 copies/mL | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Schmaldienst, MD, Study Chair — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria, Austria

REFERENCES:
- [Background] Humar A, Michaels M; AST ID Working Group on Infectious Disease Monitoring. American Society of Transplantation recommendations for screening, monitoring and reporting of infectious complications in immunosuppression trials in recipients of organ transplantation. Am J Transplant. 2006 Feb;6(2):262-74. doi: 10.1111/j.1600-6143.2005.01207.x. PMID 16426310
- [Background] Benichou C. Criteria of drug-induced liver disorders. Report of an international consensus meeting. J Hepatol. 1990 Sep;11(2):272-6. doi: 10.1016/0168-8278(90)90124-a. PMID 2254635
- [Background] Kasiske BL, Vazquez MA, Harmon WE, Brown RS, Danovitch GM, Gaston RS, Roth D, Scandling JD, Singer GG. Recommendations for the outpatient surveillance of renal transplant recipients. American Society of Transplantation. J Am Soc Nephrol. 2000 Oct;11 Suppl 15:S1-86. PMID 11044969